CLINICAL TRIAL: NCT01520844
Title: Multicentric Cohort of HIV Patient With Extrem Profil
Brief Title: the ANRS CO21 " Extreme " Cohort (CODEX)
Acronym: CODEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ANRS CO21 CODEX
Record Dates: First submitted 2011-08-09; First posted 2012-01-30 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort study (Other): Blood sampling
  Interventions: Biological: blood sampling

INTERVENTIONS:
Biological: blood sampling — blood sampling

SUMMARY:
A consortium of research teams has studied the immunovirological characteristics of these patients:

The ANRS CO15 ALT cohort The ANRS CO18 HIV Controller cohort the ANRS EP47 VISCONTI study

DETAILED DESCRIPTION:
Two cohorts of patients with a phenotype of HIV resistance exist in France. The ANRS CO15 ALT cohort was set up in 1994. 71 patients were enrolled defined on immunological criteria: CD4 T cell count above 600/mm3 with a stable or increasing count (positive or zero slopes) on at least three consecutive exams performed during the last 5 years whatever the viral load was, with a known HIV infection for at least 8 years. A consortium of research teams has studied the immunovirological characteristics of these patients. After 16 years of follow-up, 6 patients are still actively followed. The main results have shown the lack of deletion in viral genes nor any functional viral defects, a small size for the viral reservoir, and distinctive genetic characteristics of the host (HLA, chemokines) which lead to potent immune cell responses associated with virus control.

The ANRS CO18 HIV Controller cohort set up in 2009 is stemming from the French National Observatory of HIV Controllers which was active between 2006 and 2008 (Study ANRS EP36). 152 patients are enrolled who are defined on virological criteria: the last 5 plasmatic viral loads should be below 400 copies/mL without any antiretroviral treatment, in HIV-infected patients for more than 5 years. A consortium of research teams has studied these patients and has shown that Controllers are infected with replication-competent HIV, that HIV infects CD4 T cells but that the viral replication in CD4 T cells is fully controlled by CD8 T cells.

In addition, the ANRS EP47 VISCONTI study identified 14 patients who had been able to maintain plasmatic viral loads below 400 copies/ml for more than 7 years in the absence of antiretroviral treatment. Differently from HIV controllers, naïve of antiretroviral treatment, the patients from the VISCONTI study started therapy within ten weeks of primary infection and kept it for a median of three years before treatment discontinuation (Post-Treatment Controllers or PTC). The initial analyses revealed important clinical and immunogenetic differences between post-treatment and natural controllers, suggesting that PTC were not naturally predispose to control infection and that they succeeded thanks to initial therapeutic intervention. The mechanisms associated with long-term control in post-treatment controllers also appear different from the main mechanisms identified in HIV controllers. The main objective now is to gather in a common cohort patients with a particular resistance to HIV infection, either with an immunological control (ALT) or a natural (HIV Controllers) or induced virological control (PTC). The enrolled patients will be the patients already enrolled in the cohorts CO15 and CO18, the ANRSEP47 VISCONTI study, and new patients. This will allow common physiopathological studies to precise the mechanisms leading to the virus control and CD4 homeostasy. A better knowledge of the mechanisms of viral control and immune response preservation is very important in the setting of vaccine perspectives and in the perspective of implementing new therapeutic interventions to induce remission of HIV infection. This cohort will allow common research projects with common funding, a better visibility both for clinicians who see patients with unusual phenotypes and for international research. Such a cohort will be unique in the world by its size and the presence of these three complementary groups of patients. The two main objectives for the " Extreme " cohort (ANRS CO21 CODEX) are clinical and immunovirological. We wish to precise the impact of a prolonged untreated HIV infection, to describe the frequency of the "immunological escapes" (CD4 T cell decrease) or "virological escapes" (permanent or transient viral load increase), and to identify predictive markers of HIV control. We wish to study the genetic characteristics of the patients and those of their viruses, the innate and adaptative immune responses directed against HIV and other viruses, the consequences of inflammation, and the characteristics of the loss of control.

ELIGIBILITY:
Inclusion Criteria:

* Patient infected with HIV-1 and not co-infected with HIV-2
* Age ≥ 18 at enrollment
* Able to give written consent
* Covered by French Social Security
* accept the constraints imposed by the study
* without antiretroviral therapy for ALT, HIC and ALT HIC groups and a control of viral load after antiretroviral treatment interruption in PTC group

ALT group: Documented HIV-1 seropositive for at least 8 years with a CD4 count above 600/mm3 with a rate stable or increasing (positive or zero slope) on at least three consecutive examinations performed during the last 5 years regardless of the viral load in the absence of antiretroviral treatment

HIC group: HIV-1 Seropositivity known for at least five years, asymptomatic, with the last 5 viral loads in HIV-RNA consecutive <400 copies / mL regardless of CD4 count in the absence of antiretroviral treatment

ALT HIC group: HIV-1 seropositive known for at least 8 years and CD4 cell counts greater than 600/mm3 with a rate stable or increasing (positive or zero slope) on at least three consecutive examinations performed during the last 5 years and with the last 5 viral loads in HIV-RNA consecutive <400 copies / mL in the absence of antiretroviral therapy.

PTC group: Patients with plasma HIV RNA > 2000 copies/mL before initiation of antiretroviral therapy. Treatment started during the primary infection (as defined by symptoms associated with seroconversion, as confirmed by a first negative ELISA and/or an incomplete P24-positive Western blot) or during the chronic phase of infection, and maintained for at least 12 months in both cases. Control of viral load after antiretroviral treatment interruption: patients must have at least two available viral load assays after stopping antiretroviral therapy. All viral loads must be <400 copies/mL for 12 months or more after stopping antiretroviral therapy, with the possible exception of one blip (one viral load above 400 copies/mL between two viral loads <400 copies/mL at least one month apart from the blip; in this case at least three viral load assays will be required). The last plasma viral load value at the time of inclusion must always be <400 copies/mL

Exclusion Criteria:

Under protection(saving) of justice

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
clinical and immuno-virological | up to 5 years

SECONDARY OUTCOMES:
mechanisms leading to the virus control and CD4 homeostasy with physiopathological studies | up to 5 years
impact of a prolonged untreated HIV infection, | up to 5 years
frequency of the "immunological escapes" (CD4 T cell decrease) or "virological escapes" (permanent or transient viral load increase) | up to 5 years
genetic characteristics of the patients and those of their viruses, the innate and adaptative immune responses directed against HIV and other viruses, the consequences of inflammation, and the characteristics of the loss of control | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lambotte, Professor, Principal Investigator — Kremlin Bicetre; Laurence Meyer, Professor, Study Chair — Methodologist INSERM CESP U1018
Locations (1):
- Lambotte, Le Kremlin-Bicêtre, France